CLINICAL TRIAL: NCT00610220
Title: Cast Versus Splint in Children With Minimally Angulated Fractures of the Distal Radius: a Randomized Controlled Trial.
Brief Title: Cast Versus Splint in Children With Acceptably Angulated Wrist Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Kathy Boutis, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000010377
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2014-05

CONDITIONS: Distal Radius Fractures
Keywords: pediatrics; wrist fractures; casting; wrist splint
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: Fiberglass short arm cast
- 2 (Experimental)
  Interventions: Device: Prefabricated wrist splint

INTERVENTIONS:
Device: Fiberglass short arm cast — Cast will be applied for a 4-week period
  Arms: 1
Device: Prefabricated wrist splint — Splint will be applied for a 4-week period
  Arms: 2

SUMMARY:
The study will compare the effectiveness of a prefabricated wrist splint with thermoplast reinforcements versus a short arm cast in skeletally immature children.

The hypothesis is that the commercially available wrist splint is at least as effective as traditional casting with respect to recovery of physical function.

DETAILED DESCRIPTION:
Acceptability angulated wrist bone fractures in children carry an excellent long-term prognosis because of the unique capacity of skeletally immature bones to heal via remodeling. Their management varies widely and there is virtually no scientific evidence supporting one treatment modality over another. Importantly, the most common treatment modality of cast application for four to six weeks is associated with many inconveniences. There are commercially available wrist splints that offer a more convenient alternative. Wrist splints likely have comparable immobilization and symptom relief, while simultaneously allowing for easier bathing and less reliance on subspeciality care. Preliminary adult evidence suggests that, in a comparable adult fracture, splinting may offer a safe alternative to casting, with earlier resumption of the usual activities. However, this treatment modality needs to be compared to the traditional casting management in the pediatric population before it can be recommended for clinical practice.

This study will be the first to challenge the current practice of routine casting and compare it to a commercially available wrist splint with respect to recovery of physical function in children with acceptably angulated wrist fractures. In addition, standardized treatment of these fractures with a splint may be associated with lower morbidity, reduced use of health care resources, and have the potential for cost savings.

This study will compare, in skeletally immature children, the functional outcomes that result from treatment with a prefabricated wrist splint versus a short arm cast in acceptably angulated distal radius fractures. Secondly, the cost-effectiveness of the splint relative to the cast will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally immature children.
2. Children must have a bone age of ≥ 5 years of age.
3. Less than or equal to 15° angulation in the sagittal plane and ≤ 0.5 cm displacement in the frontal plane.

Therefore, all skeletally immature children ≥ 5 years and with a bone age of ≤ 11 years who present to the ED of HSC with acute distal metaphyseal radius +/- ulnar fractures that meet criteria for acceptable angulation and displacement will be eligible for enrollment.

Exclusion Criteria:

1. Age < 5 years or > 12
2. The following diagnoses of distal radius fracture: buckle fracture, growth plate fractures of any kind, distal radius metaphyseal fractures with greater than 15° of angulation in the sagittal plane and/or more than 0.5 cm of displacement in the frontal plane.
3. All open fractures which require a surgical debridement.
4. All children at risk for pathological fractures such as those with congenital or acquired generalized bony disease. Stricter immobilization and a different prognosis may be applicable to this population.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Modified performance Activities Scale for Kids (ASKp) score | 6 weeks

SECONDARY OUTCOMES:
Changes in Angulation and/or displacement | 1 and 4 weeks
Pain | 1 and 4 weeks
Duration of immobilization device | 1 and 4 week follow-up visits
Grip Strength | 6 week follow-up visit
Range of Motion | Week 6
Patient Preference for their Device | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Boutis, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Boutis K, Willan A, Babyn P, Goeree R, Howard A. Cast versus splint in children with minimally angulated fractures of the distal radius: a randomized controlled trial. CMAJ. 2010 Oct 5;182(14):1507-12. doi: 10.1503/cmaj.100119. Epub 2010 Sep 7. PMID 20823169